CLINICAL TRIAL: NCT00025896
Title: A Prospective Multinational, Multicenter, Clinical Trial of the Safety and Efficacy of Recombinant Human Acid Alpha-Glucosidase (rhGAA) in Cross-Reacting Immunologic Material-Positive Patients With Classical Infantile Pompe Disease
Brief Title: Safety and Efficacy of Recombinant Human Acid Alpha-Glucosidase in the Treatment of Classical Infantile Pompe Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGLU-001-00
Record Dates: First submitted 2001-10-31; First posted 2001-11-01 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Pompe Disease; Glycogen Storage Disease Type II; Acid Maltase Deficiency Disease; Glycogenosis 2
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — GAA protein, human

INTERVENTIONS:
Drug: recombinant human acid alpha-glucosidase (rhGAA)

SUMMARY:
Pompe disease is caused by a deficiency of a critical enzyme in the body called acid alpha glucosidase (GAA). Normally, GAA is used by the body's cells to break down glycogen (a stored form of sugar) within specialized structures called lysosomes. In infants with severe cases of Pompe disease (called Classical Infantile Pompe disease), an excessive amount of glycogen accumulates and is stored in various tissues, especially heart, skeletal muscle, and liver, which prevents their normal function. This study being conducted to evaluate the safety and effectiveness of recombinant human acid alpha-glucosidase (rhGAA) as a potential enzyme replacement therapy for Pompe disease. Patients diagnosed with Classical Infantile Pompe disease who have a small, but inactive, amount of natural GAA enzyme present in their bodies (called Cross-Reacting Immunologic Material-Positive or "CRIM (+)" patients), will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Classical Infantile Pompe Disease
* endogenous GAA activity < 1.0%
* cardiomegaly
* cardiomyopathy
* CRIM (+)
* ability to comply with the clinical protocol which will require extensive clinical evaluations

Exclusion Criteria:

* respiratory insufficiency
* cardiac failure
* major congenital abnormality
* any other medical condition that could potentially decrease survival
* CRIM (-)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8
Dates: Start 2001-05; Study Completion 2002-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Kishnani PS, Goldenberg PC, DeArmey SL, Heller J, Benjamin D, Young S, Bali D, Smith SA, Li JS, Mandel H, Koeberl D, Rosenberg A, Chen YT. Cross-reactive immunologic material status affects treatment outcomes in Pompe disease infants. Mol Genet Metab. 2010 Jan;99(1):26-33. doi: 10.1016/j.ymgme.2009.08.003. PMID 19775921